CLINICAL TRIAL: NCT00446875
Title: Efficacy of Oral Sucrose and Maternal Contact During Routine Immunizations in Postnatal Infants
Brief Title: Analgesic Properties of Oral Sucrose During Immunizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SeedHatfield
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Procedural Pain
Keywords: Pain; Procedural pain; Sucrose; Infant
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind (subject, Investigator)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucrose (Experimental): Participants received oral sucrose (0.6mL/Kg) 2 minutes prior to the combind DTaP, IPV, and Hep B (Hib and PCV7) vaccine.
  Interventions: Other: Administration of oral Sucrose
- Placebo (Placebo Comparator): Participants received Placebo (sterile water, 0.6mL/Kg) 2 minutes prior to the combind DTaP, IPV, and Hep B (Hib and PCV7) vaccine.
  Interventions: Other: Administration of oral Placebo

INTERVENTIONS:
Other: Administration of oral Sucrose — Participants received oral sucrose 2 minutes prior to the combind DTaP, IPV, and Hep B vaccine.
  Arms: Sucrose
Other: Administration of oral Placebo — Participants received Placebo 2 minutes prior to the combind DTaP, IPV, and Hep B vaccine.
  Other Names: sterile water
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the analgesic properties of oral sucrose during routine immunizations. Hypothesis: Oral sucrose solution and maternal contact will significantly decrease the objective measures of acute pain during routine immunizations.

DETAILED DESCRIPTION:
The purpose of this study is to examine the analgesic properties of oral sucrose during routine immunizations. Hypothesis: Oral sucrose solution and maternal contact will significantly decrease the objective measures of acute pain during routine immunizations.

Acute pain during early life may alter infant pain responses, cognitive development and behavioral outcomes. Infants respond to immunizations with significant pain and distress. This study will examine the analgesic properties of oral sucrose and maternal holding in postnatal infants.

Comparison: Administration of oral sucrose, sterile water and maternal contact 2 minutes before routine immunizations.

ELIGIBILITY:
Inclusion Criteria:

1. Currently between 4 and 11 months of age;
2. Between 37 and 42 weeks' completed gestation at birth;
3. Birth weight greater than 2.5 kg; and
4. No evidence of acute or chronic disease

Exclusion Criteria:

1. Fed 30 minutes prior to immunization;
2. Received analgesic/sedative the day of the immunizations;
3. Parent wishes to feed the infant during the immunizations;
4. Infant is diagnosed with a major congenital disorder where the behavioral responses to painful stimuli may be altered; or
5. Language barriers preclude the process of obtaining parental consent.

Ages: 3 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05-19 (Actual); Study Completion 2008-05-19 (Actual)

PRIMARY OUTCOMES:
Behavioral pain response | Baseline, and then at 2 and 5 minutes post DTaP, IPV, and Hep B vaccine
  Infants will be evaluated based on the University of Wisconsin Children's Hospital Pain Scale to score an infant's pain. Possible scores range from 0 (no pain) to 5 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Hatfield, PhD, Principal Investigator — The Penn State University
Locations (1):
- University Pediatric Associates, Penn State Children's Hospital, Hershey, Pennsylvania, United States